CLINICAL TRIAL: NCT03752775
Title: Mobile Electromyography (EMG)-Driven Exoneuromusculoskeleton for Upper Limb Rehabilitation After Stroke
Brief Title: Exoneuromusculoskeleton for Upper Limb Rehabilitation After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Xiaoling Hu, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITS/073/16
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Upper Limb Rehabilitation
Keywords: stroke; upper limb; Joint coordination
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The device assisted treatment will be administrated to patients with subacute stroke and chronic stroke. The subacute stroke group will be compared in parallel with a control group receive the conventional physical and occupational therapies.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- subacute device assisted group (Experimental)
  Interventions: Device: Robot assisted upper limb rehabilitation
- subacute conventional group (Active Comparator)
  Interventions: Device: Robot assisted upper limb rehabilitation
- chronic device assisted group (Other)
  Interventions: Device: Robot assisted upper limb rehabilitation

INTERVENTIONS:
Device: Robot assisted upper limb rehabilitation — The patients in the experimental and the other arms will receive 20 session device assisted upper limb rehabilitation. In each session, a subject will conduct multi-joint coordinated upper limb motions for 1 hour.

SUMMARY:
A new clothing robotic arm was developed for multi-joint coordinated upper limb rehabilitation after stroke. Patients after stroke will be recruited to evaluate the rehabilitation effectiveness of the device assisted upper limb rehabilitation. Both patients with chronic stroke and subacute stroke will be investigated.

DETAILED DESCRIPTION:
A new robotic arm, named mobile exo-neuro-musculo-skeleton, was developed for upper limb rehabilitation. The system integrated the advantages of exoskeleton, soft robot, and neuromuscular electrical stimulation. It is noninvasive, light in weight, comfortable to wear, and can support the motions at the elbow, the wrist and the fingers. The device is a mobile system interfaced with a mobile app by a user.

The device assisted upper limb rehabilitation will be applied to inpatients with subacute stroke. The rehabilitation effects on the motor restoration in the upper limb will be compared with the conventional physical and occupational therapies. The rehabilitation effects of the device assisted training also will be evaluated on patients with chronic stroke. The motor improvements after training will be investigated by comparing the pre- and post- clinical assessments. It is hypothesized that the device assisted upper limb rehabilitation will be effective in both subacute and chronic patients.

ELIGIBILITY:
Inclusion Criteria:

For the subacute groups:

* Two weeks after the onset of stroke, however less than 0.5 year
* Mini-Mental State Examination (MMSE)>21
* Able to sit up for at least 1 hour
* Fugl-Meyer Assessment (FMA) upper limb <30
* Modified Ashworth Score (MAS) at the elbow, wrist and fingers <3
* Detectable EMG on the target driving muscles (i.e., 3 times of the standard deviation above the baseline)

For the chronic device assisted group:

* At least 0.5 year after the onset of stroke
* Mini-Mental State Examination (MMSE)>21
* Able to sit up for at least 1 hour
* Fugl-Meyer Assessment (FMA) upper limb <30
* Modified Ashworth Score (MAS) at the elbow, wrist and fingers <3
* Detectable EMG on the target driving muscles (i.e., 3 times of the standard deviation above the baseline)

Exclusion Criteria:

Subjects will be excluded if they do not meet the above inclusion criteria, or had the following conditions:

* Currently pregnant
* Dysphasia (language deficiency)
* Post-stroke neglect
* Pacemaker implantation,
* Involved in drug studies, other clinical trials, or concurrent medication/occupational/physical treatments on the upper limb
* The overall medical condition not suitable for the training (e.g., severe cardiac problem, unstable blood pressure, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) of the Upper Limb before the training | For each subject, the FMA score will be measured one day before the training.
Fugl-Meyer Assessment (FMA) of the Upper Limb after the training | For each subject, the FMA score will be measured one day after the 20-session training program.
Fugl-Meyer Assessment (FMA) of the Upper Limb 3-month follow-up | For each subject, the FMA score will be measured 3 months later after the last day of the training.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | For each subject, the MAS score will be measure one day before the training, one day after the 20-session training program, and 3 months later after the last day of the training.
Action Research Arm Test (ARAT) | For each subject, the ARAT score will be measure one day before the training, one day after the 20-session training program, and 3 months later after the last day of the training.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nam C, Zhang B, Chow T, Ye F, Huang Y, Guo Z, Li W, Rong W, Hu X, Poon W. Home-based self-help telerehabilitation of the upper limb assisted by an electromyography-driven wrist/hand exoneuromusculoskeleton after stroke. J Neuroeng Rehabil. 2021 Sep 15;18(1):137. doi: 10.1186/s12984-021-00930-3. PMID 34526058
- [Derived] Nam C, Rong W, Li W, Cheung C, Ngai W, Cheung T, Pang M, Li L, Hu J, Wai H, Hu X. An Exoneuromusculoskeleton for Self-Help Upper Limb Rehabilitation After Stroke. Soft Robot. 2022 Feb;9(1):14-35. doi: 10.1089/soro.2020.0090. Epub 2020 Dec 3. PMID 33271057